CLINICAL TRIAL: NCT02901535
Title: Tele-spirometry in Primary Care - Randomized Clinical Trial Cluster: the Effectiveness of Multifaceted Intervention in Symptoms Patients With Respiratory Illness
Brief Title: Tele-spirometry in Primary Care-Randomized Clinical Trial Cluster:Telemedicine in Chronic Obstructive Pulmonary Disease
Acronym: RESPIRANET-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 227190 COPD
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: telemedicine; chronic obstructive pulmonary disease; Primary Health care; spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Remote Consultation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Spirometry in baseline Spirometry - 20 weeks
  Interventions: Other: Spirometry; Other: Spirometry - 20 weeks
- Intervention (Experimental): Spirometry in baseline Teleconsultation Telemonitoring Spirometry - 20 weeks
  Interventions: Other: Spirometry; Other: telemonitoring; Other: teleconsultation; Other: Spirometry - 20 weeks

INTERVENTIONS:
Other: Spirometry — Spirometry in baseline
Other: telemonitoring — telemonitoring (phone call nurse - 45 and 90 days)
  Arms: Intervention
Other: teleconsultation — teleconsultation (general practioner received phone call to respiratory care)
  Arms: Intervention
Other: Spirometry - 20 weeks — Spirometry (20 weeks)

SUMMARY:
The purpose of this study is to determine the effectiveness of telemedicine multifaceted intervention in symptoms patients with chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
This study is a randomized clinical trial for patients with chronic obstructive pulmonary disease from a primary care. The purpose is to determine the effectiveness of telemedicine (teleconsultation and telemonitoring) in control of chronic obstructive pulmonary disease symptoms.

ELIGIBILITY:
Inclusion Criteria:

* spirometry from TelessaudeRS-Universidade Federal do Rio Grande do Sul (from randomization cluster), Modified Medical Research Council Dyspnea > 0

Exclusion Criteria:

* normal or restrictive spirometry, low quality spirometries (inadequate)

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms | 20 a 22 weeks
  Modified Medical Research Council Dyspnea Scale (difference in mMRC)

SECONDARY OUTCOMES:
Spirometry - FEV1 | 20 a 22 weeks
  spirometry parameters - FEV 1 (forced expiratory volume in one second)
Spirometry - FVC | 20 a 22 weeks
  spirometry parameters - FVC (forced vital capacity)

CONTACTS AND LOCATIONS:
Overall Officials: Erno Harzheim, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- TelessaudeRS-Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided